CLINICAL TRIAL: NCT06380673
Title: Stepwise Heat-Denaturated Protein Introduction for Tolerance Induction in Food Allergy
Acronym: TEHITI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, Clinic Head in Pediatrics-Allergy at UZ Leuven, Head of the Allergy and Clinical Immunology Research group at KU Leuven (prof., dr.), Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: s68299
Record Dates: First submitted 2024-03-19; First posted 2024-04-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Food Allergy; Cow Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stepwise introduction using gradually shorter heating of cow's milk proteins (Other): Step 1: open introduction of 20' cooked cow's milk (at least 10 mL per portion, 2-3X a week) for 3 months.
  Step 2: open introduction of 15' cooked cow's milk (at least 10 mL per portion, 2-3X a week) for 3 months.
  Step 3: open introduction of 10' cooked cow's milk (at least 10 mL per portion, 2-3X a week) for 3 months.
  Step 4: open introduction of 5' cooked cow's milk (at least 10 mL per portion, 2-3X a week) for 3 months.
  Interventions: Other: Implementation of cow's milk in decreasingly heated forms
- Stepwise introduction using the Flemish Milk Ladder (Other): The first 5 steps of the Flemish Milk Ladder (each containing a, b and c part) will be gradually introduced at home, each step for 21 days (2-3X a week during 3 consecutive weeks after which 3 days "rest"). We consider the 6th step the equivalent of tolerance induction so step 6 will be allowed once the OFC with uncooked milk is passed.
  Interventions: Other: Implementation of cow's milk in decreasingly heated forms
- Control arm with introduction of 20' cooked cow's milk (Other): Step 1: open introduction of 20' cooked cow's milk (at least 10 mL per portion, 2-3X a week) for 12 months.
  Interventions: Other: Implementation of heated cow's milk
- Healthy age-matched subjects (Other): For work package 2, 15 healthy age-matched subjects are included to compare immunological mechanisms with.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Implementation of cow's milk in decreasingly heated forms — Implementation of cow's milk in decreasingly heated forms in cow's milk allergic subjects, tolerant to heated cow's milk, to assess the influence on tolerance induction.
  Arms: Stepwise introduction using gradually shorter heating of cow's milk proteins; Stepwise introduction using the Flemish Milk Ladder
Other: Implementation of heated cow's milk — Implementation of heated cow's milk in cow's milk allergic subjects, tolerant to heated cow's milk, to assess the influence on tolerance induction.
  Arms: Control arm with introduction of 20' cooked cow's milk
Other: No intervention — Healthy subjects undergo no intervention.
  Arms: Healthy age-matched subjects

SUMMARY:
This interventional study aims to validate an early heated protein introduction protocol in cow's milk allergic children who already developed tolerance towards extensively heated cow's milk, in order to speed up the development of complete cow's milk tolerance. Natural complete tolerance induction towards cow's milk takes several years of strict cow's milk avoidance with high risk of anaphylaxis by accidental cow's milk intake. By shortening the time towards complete tolerance, not only the quality of life of both children and parents ameliorates drastically, the time frame for potential anaphylactic reactions is also strongly reduced and can be considered as a preventive strategy to reduce allergic reactions too. Moreover, this strategy has proved efficient for hen's egg allergy. The main question this study wants to answer is whether a 12 months stepwise heated cow's milk introduction (either by gradual reduction of the cooking time or by the use of the Flemish Milk Ladder) in 20'-cooked cow's milk tolerant subjects, results in a larger proportion of complete cow's milk tolerant children after 12 months compared to natural tolerance induction (with 20' cooked milk introduction only).

DETAILED DESCRIPTION:
WP 1: Gradual introduction of less heated cow's milk proteins in 20'-cooked cow's milk tolerant children.

When inclusion criteria are met and informed consent from the parents (and when old enough, assent from the children) is obtained, children will be included in the trial. During the inclusion visit an open 20' cooked milk oral food challenge (OFC) needs to be passed in the hospital. Each visit a validated pedQuality of life (QoL) questionnaire will be taken and blood will be drawn to determine baseline specific IgE (sIgE) and IgG4 to cow's milk. Subjects (n=75) are randomized in a 1/1/1 ratio across three arms for 12 months to study the arm's tolerance inducing capacity (see Arms and Interventions for more information). After 6 months patients are invited for an intermediate visit. After 12 months, a OFC with unheated milk will be performed in all children during their challenge visits. Three months after the OFC, the children will be invited for a termination visit. Children who did not pass the OFC with unheated cow's milk after 12 months, will be invited to an observational 48 months follow-up study, in order to later-on retrieve the potential moment of complete cow's milk tolerance induction by clinical files.

WP2: Study of the immunological mechanisms (Treg and Breg induction and switch to IgG4-producing B cells).

Venous blood will be taken from all 75 children recruited for WP1 at enrolment and at the challenge and termination visit and from 15 healthy age-matched children, after obtaining children's oral or written assent (where appropriate) and parent's informed consent. Peripheral blood mononuclear cells (PBMCs) will be isolated and stimulated by cow's milk proteins as well as a positive control. Membrane markers associated with regulatory activity on T cells will be studied by flow cytometry (FC), as well as cytokine production in the supernatant by meso scale discovery. Furthermore, B cells will be studied after PBMC stimulation by FC. Cow's milk specific IgG4 and cytokine production will also be studied in this culture supernatant.

WP3: In vitro BATs to mimic the outcome of OFC.

In vitro Basophil activation tests (BATs) will be fine-tuned by preparing extracts for 20', 15', 10', 5' cooked and fresh cow's milk. Fine-tuning will include the comparison of new protein extract batches with the first batches, the absence of background basophil activation upon contact with the lowest dose of allergen extract and the comparison of basophil activation of healthy and of allergic children in different phases of cow's milk tolerance, who should show differences depending on the grade of tolerance. After fine-tuning, BATs will be performed as described above with 3 (or 5) extracts from cow's milk at baseline, challenge visit and termination visit in all children recruited within the study.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-18y) had or have a clinical diagnosis of IgE mediated cow's milk allergy based on positive history as well as skin prick testing and/or specific IgE detection by CAPtest in an allergy clinic.
* Children are at least 12 months old before introduction of heated cow's milk is considered.
* Children did not suffer from grade 4 anaphylaxis due to cow's milk-ingestion at presentation.
* Children have specific IgE levels to Bos d 8 below 1.2 kU/mL and/or children passed 20' cooked cow's milk provocation test executed on clinical judgement.

Exclusion Criteria:

* Children had grade 4 anaphylaxis due to cow's milk ingestion.
* Children are younger than 12 months old at the moment of passing 20' cooked cow's milk OFC.
* Parents are not able or not willing to adhere to a specific cow's milk protein-containing diet on a regular basis at home.
* Multiple food allergy, not compatible with any of the choices in the Flemish Milk Ladder.
* Parents and/or children are not willing to give IC/assent.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete cow's milk tolerance after 12 months of stepwise heated cow's milk introduction | 12 months
  We here want to test the hypothesis that a total period of 12 months stepwise heated cow's milk introduction (either by gradual reduction of the cooking time or by the use of the Flemish Milk Ladder) in 20'-cooked cow's milk tolerant subjects, results in a larger proportion of complete cow's milk tolerant children after 12 months compared to natural tolerance induction (with 20' cooked milk introduction only).

SECONDARY OUTCOMES:
Time to complete tolerance in all three arms | 12 months
  We will study how long it takes for the subjects of each arm to develop complete tolerance toward cow's milk.
Quality of life in all three arms | 12 months
  We will compare Quality of life (QoL) in each arm by comparing the questionnaires filled out by subjects and their parents in each arm.
Clinical reactions | 12 months
  We will compare the presence of clinical reactions after food introduction at home in each arm. Clinical reactions could be anaphylaxis, rhinitis, atopic dermatitis and so forth.
Side effects | 12 months
  We will compare the presence of side effects after food introduction at home in each arm. Side effects could be development of unpleasant taste, refusal of other food, development of eosinophilic esophagitis and so forth.
IL-10-producing cow's milk specific regulatory T and B cells | Three times in 12 months
  We will study the induction of IL-10-producing cow's milk specific Treg cells and Breg cells in vitro paralleling tolerance induction. Blood samples are drawn at enrolment, at challenge and termination visit.
BATs to mimic the outcome of cow's milk provocation tests | Three times in 12 months
  We will study whether we can correlate the results of the in-house developed in vitro Basophil activation tests (BAT) with different heated cow's milk-containing extracts to the results of the cow's milk provocation test after 12 months. Blood samples are drawn at enrolment, at challenge and termination visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Leus, MD, Principal Investigator — Maria Middelares Hospital, Gent; Katrien Coppens, MD, Principal Investigator — Imelda Hospital, Bonheiden; Sophie Verelst, MD, Principal Investigator — KU Leuven and Jessa Hospital, Hasselt; Kate Sauer, MD, Principal Investigator — AZ Sint-Jan AV
Locations (5):
- Belgium (5):
  - Imelda Hospital Bonheiden, Bonheiden
  - AZ Sint-Jan, Bruges
  - AZ Maria Middelares, Ghent
  - Jessa Hospital, Hasselt
  - UZ Leuven Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: No